CLINICAL TRIAL: NCT04042688
Title: Intra-articular Administration of 3.0g Tranexamic Acid Has no Effect on Reducing Intra-articular Hemarthrosis and Postoperative Pain After Primary Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hoon Bae, Associate Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GR0011
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Patients were randomly allocated to one of two groups during preoperative preparation by computer-generated randomization. Treatment group; IA administration of TXA, control group; no TXA administration
  Interventions: Drug: intraarticular administration of tranexamic acid
- Control gorup (No Intervention)

INTERVENTIONS:
Drug: intraarticular administration of tranexamic acid — Intraarticular administration with concentration of 30mg/mL was selected. The operation room nurses prepared 3g tranexamic acid in 100 mL of saline solution during operation. After finishing surgical wound suture and orthopaedic surgeons related to this study left operation room, the orthopaedic residents who were not involved in the postoperative evaluation administered tranexamic acid solution through suprapatellar pouch before tourniquet release in patients in the treatment group. The control group did not receive any solution. intraarticular drain was not inserted in all patients.
  Arms: Treatment group

SUMMARY:
The purpose of this study was to investigate whether intraarticular administration of tranexamic acid could reduce hemarthrosis and postoperative pain in patients following anterior cruciate ligament reconstruction. The hypothesis of the study was that patients treated with intraarticular tranexamic acid would have significantly less postoperative hemarthrosis and less pain in the early phase of the rehabilitation process compared with those without intraarticular tranexamic acid .

DETAILED DESCRIPTION:
Intervention Based on the previous studies, intraarticular administration with concentration of 30mg/mL was selected. The operation room nurses prepared 3g tranexamic acid in 100 mL of saline solution during operation. After finishing surgical wound suture and orthopaedic surgeons related to this study left operation room, the orthopaedic residents who were not involved in the postoperative evaluation administered tranexamic acid solution through suprapatellar pouch before tourniquet release in patients in the treatment group. The control group did not receive any solution. intraarticular drain was not inserted in all patients.

Outcome Demographic variables (age, sex, body mass index, and time from injury to surgery), clinical outcomes and surgical records including operative time, bleeding amounts, meniscus and cartilage lesions were collected by an independent orthopaedic resident. Primary outcome was a blood loss calculated based on hemoglobin balance. We assumed that blood volume in ml on the second day after surgery was the same as that before surgery. Blood volume was estimated according to the method of Nadler and colleagues taking sex, body mass and height into account. The loss of Hemoglobin was then estimated according to the formula.

Hemoglobin loss=Blood volume*(Hemoglobin concentration before surgery - Hemoglobin concentration after surgery)*0.001+total amount of allogenic hemoglobin transfused

The secondary outcome was an extent of pain measured by a visual analog scale at a consistent time in the afternoon of postoperative day 1 (PD 1) and for the next 4 day.The pain visual analog scale is a numeric response on a scale from 0 to 10, with 0 denoting no pain and 10 signifying severe pain. The other secondary outcomes included mid-patellar circumference at postoperative day 2 and day 5 and knee range of motion after 6 weeks from operation, which were measured by an independent orthopaedic fellow. The patellar circumference was measured transverse axis of the patella center to evaluate intra-articular effusion. To minimize inter-observer variance of the patellar circumference, we considered the difference between the preoperative and the postoperative results. The range of motion was documented as the extension and flexion degrees using an orthopaedic goniometer.

ELIGIBILITY:
Inclusion Criteria:

* primary single bundle anterior cruciate ligament reconstruction using a hamstring autograft with or without meniscus surgeries

Exclusion Criteria:

* use of other grafts (allograft, bone patellar tendon bone autograft)
* revision anterior cruciate ligament reconstruction,
* concomitant knee cartilage or collateral ligament surgeries
* history of knee surgery on affected knee
* concomitant fracture
* significnat preoperative pain (Visual analoge score >5)
* coagulation or bleeding disorders
* preoperative anticoagulation treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
blood loss | 2 days
  Primary outcome was a blood loss calculated based on hemoglobin balance. We assumed that blood volume in ml on the second day after surgery was the same as that before surgery. Blood volume was estimated according to the method of Nadler and colleagues taking sex, body mass and height into account. The loss of Hemoglobin was then estimated according to the formula.
  Hemoglobin loss=Blood volume*(Hemoglobin concentration before surgery - Hemoglobin concentration after surgery)*0.001+total amount of allogenic hemoglobin transfused.

SECONDARY OUTCOMES:
extent of pain | 1 day and 5days
  The secondary outcome was an extent of pain measured by a visual analog scale at a consistent time in the afternoon of postoperative day 1 and for the next 4 day.The pain visual analog scale is a numeric response on a scale from 0 to 10, with 0 denoting no pain and 10 signifying severe pain.
patellar circumference | 2days and 5days
  The patellar circumference was measured transverse axis of the patella center to evaluate intra-articular effusion
range of motion | 6 weeks
  The range of motion was documented as the extension and flexion degrees using an orthopaedic goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Jihoon Bae, Principal Investigator — Department of Orthopaedic Surgery at Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JW, Kim SG, Kim SH, Cho HW, Bae JH. Intra-articular Administration of Tranexamic Acid Has No Effect in Reducing Intra-articular Hemarthrosis and Postoperative Pain After Primary ACL Reconstruction Using a Quadruple Hamstring Graft: A Randomized Controlled Trial. Orthop J Sports Med. 2020 Jul 22;8(7):2325967120933135. doi: 10.1177/2325967120933135. eCollection 2020 Jul. PMID 32743011